CLINICAL TRIAL: NCT03521791
Title: Efficacy and Safety of PRO-155 (Zebesten Ofteno®) on Inflammation of the Conjunctival Surface in Subjects With Grade I-III Pterygium vs Placebo.
Brief Title: Efficacy and Safety of PRO-155 on Inflammation of the Conjunctival Surface in Subjects With Grade I-III Pterygium vs Placebo.
Acronym: PRO-155/IV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOPH155-0415/IV
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Pterygium; Ocular Pain; Ocular Inflammation; Post-surgical Inflammation
Keywords: zebesten; ocular anti-inflammatory; ocular analgesic; pterygium; anti-inflammatory non-steroidal ophthalmic
MeSH Terms: conditions — Pterygium; Eye Pain | interventions — bromfenac

STUDY DESIGN:
Intervention Model Description: A controlled, randomized, double-blind, masked clinical trial comparing the safety and efficacy of PRO-155 in the treatment of conjunctival hyperemia in pterygium I to III compared to placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The double-blind study is a procedure in which the subject and the principal investigator do not know which of the intervention groups was assigned to the subject of the study. To achieve the blinding of the drug, both the investigational drug and the placebo, will be packed in the same bottle, containing the same legends on the label. The blinding codes are protected by a person outside the study designated by the sponsor. The codes are also available in the research center (fully sealed), so that they can be consulted by the Investigator in the event that the subject presents a serious adverse event, prior authorization of the study sponsor, as well as strict continuous blindness during the analysis of data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-155 (Experimental): Pro-155: 1 drop 2 times a day in the period of vigil in the conjunctival cul-de-sac for 20 days
  Interventions: Drug: PRO-155
- Placebo (Placebo Comparator): Placebo 1 drop 2 times a day in the period of vigil in the conjunctival cul-de-sac
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRO-155 — PRO-155 (Zebesten ofteno®) Active agent: bromfenac 0.90 mg / mL, dropper bottle of low density polyethylene for multidose administration in the form of an ophthalmic solution of 5 mL (milliliters). Sanitary registry in Mexico: 108M2014
  Sodium hyaluronate 0.4% [Lagricel ofteno®] 1 drop 3 times a day in the period of vigil in the conjunctival cul-de-sac
  Other Names: zebesten; bromfenac
  Arms: PRO-155
Other: Placebo — The placebo is constituted by agents, additives and vehicles, of the formulation PRO-155 without pharmacological activity. It is dispensed in dropper bottle of low density polyethylene for multi-dose administration in the form of ophthalmic solution of 5 mL
  Sodium hyaluronate 0.4% (Lagricel ofteno®) 1 drop 3 times a day in the period of vigil in the conjunctival cul-de-sac
  Arms: Placebo

SUMMARY:
Title of the study Efficacy and safety of PRO-155 (Zebesten ofteno®) on inflammation of the conjunctival surface in subjects with grade I-III pterygium vs placebo.

Hypothesis H0. The Zebesten® ophthalmic solution (bromfenac 0.09%) is less effective and safe than placebo in reducing conjunctival hyperemia in subjects with grade I-III pterygium.

H1 The Zebesten® ophthalmic solution (bromfenac 0.09%) is more effective and safe than placebo in reducing conjunctival hyperemia in subjects with grade I-III pterygium.

Objective

To evaluate the efficacy and safety of PRO-155 (bromfenac 009%) ophthalmic solution in the treatment of conjunctival hyperemia and ocular surface inflammation in a clinical model of pterygium grade I to III.

DETAILED DESCRIPTION:
Variables to be evaluated Visual ability Intraocular pressure. Ocular surface Exploration of the previous segment. Exploration of the posterior segment. Lacrimal rupture time. Corneal de-epithelialization Conjunctival de-epithelialization Adverse events.

PHARMACOLOGICAL INTERVENTION

The pharmacological intervention will consist of the instillation of the ophthalmological solution in the conjunctival cul-de-sac, during the waking period, to any of the following study groups:

* Group 1:

  * Sodium hyaluronate 0.4% [Lagricel ofteno®] 1 drop 3 times a day in the period of vigil in the conjunctival sac fund (the following application scheme is suggested: start: 7:00 ± 1 hours, continuation: 15:00 ± 1 hour and term: at 19:00 ± 1 hours) for 20 days
  * Pro-155 1 drop 2 times a day in the period of vigil in the conjunctival cul-de-sac (the following application scheme is recommended: start: 7:15 ± 1 hours and term: at 19:15 ± 1 hours) during 20 days
* Group 2:

  * Sodium hyaluronate 0.4% [Lagricel ofteno®] 1 drop 3 times a day in the period of vigil in the conjunctival sac fund (the following application scheme is suggested: start: 7:00 ± 1 hours, continuation: 15:00 ± 1 hour and term: at 19:00 ± 1 hours) for 20 days
  * Placebo 1 drop 2 times a day in the period of vigil in the conjunctival cul-de-sac (the following application scheme is recommended: start: 7:15 ± 1 hours and term: at 19:15 ± 1 hours) for 20 days

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 90 years.
* Both genders.
* Clinical diagnosis of grade I to III pterygium (temporal, nasal, or bitemporal).
* Possibility of going to the revisions when indicated.

Exclusion Criteria:

* Subjects with topical or systemic medication that interfere decisively in the results of the study; such as topical immunomodulators, NSAIDs, antihistamines, corticosteroids, artificial tears with conservative, vasoconstrictors etc.
* Subjects (female) with active sexual life who do not use a contraceptive method.
* Subjects of the female sex in a pregnant state or who are breastfeeding.
* Subjects of the female sex with pregnancy test in positive urine.
* Positive substance abuse
* Subjects who have participated in any clinical research study in the last 40 days.
* Subjects legally or mentally incapacitated to give their informed consent for their participation in this study.
* Subjects that can not comply with the appointments or with all the requirements of the Protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (3):
- Mexico (3):
  - catarata y glaucoma de occidente S.A de C.V., Guadalajara, Jalisco
  - Novam y Vita, Guadalajara, Jalisco
  - Consultorio PRivado Miguel Angel Villanueva, Mexico City

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-155: Pro-155: 1 drop 2 times a day in the period of vigil in the conjunctival cul-de-sac for 20 days
  PRO-155: PRO-155 (Zebesten ofteno®) Active agent: bromfenac 0.90 mg / mL, dropper bottle of low density polyethylene for multidose administration in the form of an ophthalmic solution of 5 mL (milliliters). Sanitary registry in Mexico: 108M2014
  Sodium hyaluronate 0.4% [Lagricel ofteno®] 1 drop 3 times a day in the period of vigil in the conjunctival cul-de-sac
- Placebo: Placebo 1 drop 2 times a day in the period of vigil in the conjunctival cul-de-sac
  Placebo: The placebo is constituted by agents, additives and vehicles, of the formulation PRO-155 without pharmacological activity. It is dispensed in dropper bottle of low density polyethylene for multi-dose administration in the form of ophthalmic solution of 5 mL
  Sodium hyaluronate 0.4% (Lagricel ofteno®) 1 drop 3 times a day in the period of vigil in the conjunctival cul-de-sac
Period: Overall Study
Arm/Group | PRO-155 | Placebo
Started | 76 | 90
Completed | 69 | 73
Not Completed | 7 | 17
Not completed — Protocol Violation | 7 | 17

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-155 | Placebo | Total
Number analyzed (Participants) | 41 | 42 | 83
Number analyzed (eyes) | 82 | 84 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (13.3) | 57.17 (14.4) | 55.51 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 41 | 42 | 83
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Hyperemia (CH)
Description: Conjunctival hyperemia will be evaluated as an ordinal variable, by direct observation and staged using the Efron scale as Normal / Very Light / Mild / Moderate / Severe. Based on this scale, the normal and mild stages are considered without pathologies or normal. Mild, moderate and severe are considered pathological.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Population: statistical analysis by protocol (PP)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
eyes
  Normal | 0 | 0
  Very mild | 39 | 29
  Mild | 25 | 36
  Moderate | 5 | 8
  Severe | 0 | 0
Statistical Analysis 1: Comparison: PRO-155; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.133, Chi-squared, Corrected

2. Primary Outcome: Breakup Time (BUT)
Description: breakup time lacrimal film is a continuous variable that will be measured in seconds, evaluating the time it takes to break it, is done by direct counting and the normality range and mayor to 10 seconds.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Population: Statistical analysis was performed by protocol (PP)
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
seconds | 8.29 (2.2) | 7.63 (2.3)
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.045, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Epithelial Defects (ED) Green Lissamine
Description: The epithelial defects will be evaluated by means of two stains, green lysine and fluorescein, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the oxford scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
eyes
  Green lissamine grade 0 | 41 | 44
  Green lissamine grade 1 | 21 | 21
  Green lissamine grade 2 | 4 | 8
  Green lissamine grade 3 | 3 | 0
  Green lissamine grade 4 | 0 | 0
  Green lissamine grade 5 | 0 | 0
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.333, Chi-squared, Corrected

4. Secondary Outcome: Intraocular Pressure (IOP)
Description: the intraocular pressure will be evaluated by means of the Goldman applanation tonometry whose unit of measurement is millimeters of mercury (mmHg), it is a continuous variable and its normality range is between 11 - 21 mmHg
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Population: the statistical analysis was carried out by protocol (PP)
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
mmHg | 12.45 (2.1) | 13.08 (1.8)
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.058, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Presence of Adverse Events (EAS)
Description: primary security variable the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent. Adverse events that are reported until the safety call to the 36th day of the study will be considered for this variable
Time Frame: will be evaluated at the end of the treatment at the final visit (day 36)
Population: The analysis of adverse events was done by intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 47 | 52
Participants | 13 | 19
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.394, Fisher Exact

6. Secondary Outcome: Visual Capacity
Description: The visual capacity variable will be reported using as a unit of measure a fraction, this is taken from a visual test with the Snellen primer, it is a Nominal type variable. where the optimal vision is 20/20.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
LogMAR | 0.043 (0.1) | 0.059 (0.2)
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.056, t-test, 2 sided

7. Secondary Outcome: Number of Eyes With Chemosis
Description: In a normal eye there is no presence of chemosis (it is a sign of irritation of the eye, in which the outer covering of the eye can look like a large blister) its presence indicates a pathological state and it will be evaluated if the subjects present it. The chemosis will be evaluated, as a nominal variable, by direct observation and it will be staged as present and absent, where the normality is that said variable is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Population: the statistical analysis was carried out by protocol (PP)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
eyes | 0 | 0

8. Secondary Outcome: Number of Eyes With Foreign Body Sensation (FBS)
Description: Foreign body sensation will be evaluated, as a nominal variable, by direct observation and it will be staged as present and absent, where the normality is that said variable is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Population: the statistical analysis was carried out by protocol (PP)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
eyes | 10 | 18
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.114, Fisher Exact

9. Secondary Outcome: Epithelial Defects (ED) Fluorescein Stain
Description: as for outcome 3
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Population: the statistical analysis was carried out by protocol (PP)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
eyes
  Fluorescein Grade 0 | 31 | 31
  Fluorescein Grade 1 | 27 | 33
  Fluorescein Grade 2 | 11 | 9
  Fluorescein Grade 3 | 0 | 0
  Fluorescein Grade 4 | 0 | 0
  Fluorescein Grade 5 | 0 | 0
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.117, Chi-squared, Corrected

10. Other Pre Specified Outcome: Number of Eyes With Ocular Burning (OB)
Description: primary tolerability variable
  Ocular burning is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.Frequency: At all times, almost at all times, 50% of the time, almost in no time, at any time. where the normality of the frequency is in no time.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 21)
Population: the statistical analysis was carried out by protocol (PP)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Placebo
Number analyzed (Participants) | 41 | 42
Number analyzed (eyes) | 69 | 73
eyes | 8 | 11
Statistical Analysis 1: Comparison: PRO-155 vs Placebo; Test type: Non-Inferiority — it is considered not inferior if the differences between the groups do not exceed 20%; p = 0.626, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded throughout the study, an average of 8 months.
Arm/Group | PRO-155 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/90
Other Adverse Events (participants affected / at risk) | 13/76 | 19/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-155 (N=76) | Placebo (N=90)
sickness (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomit (Gastrointestinal disorders) | 0 (0) | 1 (1)
photophobia (Eye disorders) | 2 (2) | 4 (4)
ocular burning (Eye disorders) | 5 (5) | 5 (5)
tearing (Eye disorders) | 0 (0) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
conjunctival hyperemia (Eye disorders) | 3 (3) | 11 (11)
ocular pain (Eye disorders) | 0 (0) | 2 (2)
Eye pruritus (Eye disorders) | 0 (0) | 3 (3)
Dry-eye feeling (Eye disorders) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 3 (3)
Stye (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
sore throat (General disorders) | 1 (1) | 0 (0)
Corneal epithelium defect (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator can not publish any information about the investigation without prior written authorization from the atrocifier

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT03521791/Prot_SAP_000.pdf